CLINICAL TRIAL: NCT02089061
Title: A Phase 1 Open-label, Single-sequence Study to Evaluate the Effect of Coadministration of BMS-919373 on the Single-dose Pharmacokinetics of Rosuvastatin and Atorvastatin in Healthy Subjects
Brief Title: Drug Interaction Statin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CV205-029
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Rosuvastatin + BMS-919373 (Experimental): Rosuvastatin 10 mg tablet orally once for Day 1 and 5
  BMS-919373: 100 mg dose on Day 4 and 30 mg dose once daily on Days 5, 6 and 7 of Microcrystalline suspension
  Interventions: Drug: BMS-919373; Drug: Rosuvastatin
- Cohort 2: Atorvastatin + BMS-919373 (Experimental): Atorvastatin 40 mg tablet once for Days 1 and 5
  BMS-919373: 100 mg dose on Day 4 and 30 mg dose once daily on Days 5, 6 and 7 of Microcrystalline suspension
  Interventions: Drug: BMS-919373; Drug: Atorvastatin

INTERVENTIONS:
Drug: BMS-919373
  Other Names: IKur Inhibitor
Drug: Rosuvastatin
  Other Names: Crestor®
  Arms: Cohort 1: Rosuvastatin + BMS-919373
Drug: Atorvastatin
  Other Names: Lipitor®
  Arms: Cohort 2: Atorvastatin + BMS-919373

SUMMARY:
This purpose of this study is to assess the effects of BMS-919373 on the single dose Pharmacokinetics (PK) of Rosuvastatin and Atorvastatin in healthy subjects.

DETAILED DESCRIPTION:
Primary Purpose: Other - To assess the effects of BMS-919373 on the single dose PK of Rosuvastatin and Atorvastatin in healthy subjects

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Signed Written Informed Consent form
* Healthy subjects as determined by no clinically significant deviation from normal in medical and surgical history, physical examination, physical measurements, vital signs, 12-lead ECG, 24-hour telemetry, and clinical laboratory tests
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive
* Men and women, ages 18 to 55 yrs, inclusive

Exclusion Criteria:

* Current or history of cardiovascular diseases, including arrhythmias, coronary heart disease, and congestive heart failure
* Current or history of symptomatic hypotension
* Current or history of liver diseases, including cirrhosis and liver failure
* Current or history of kidney diseases, including nephrotic syndrome, renal failure, nephrolithiasis, and urolithiasis
* Current or history of neurological diseases, including presyncope, syncope, convulsive disorders such as epilepsy, cerebral thrombosis and cerebral embolism, transient ischemic attack, and stroke; or mental disorders Exceptions for presyncope/syncope related to vasovagal responses are allowable at the discretion of the investigator
* History of significant head injury in the last 2 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Rosuvastatin and Atorvastatin | 28 timepoints up to day 10
Area under the plasma concentration-time curve from time zero to 72 hours (AUC(0-72)) of Rosuvastatin and Atorvastatin | 26 timepoints up to day 8
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of Rosuvastatin and Atorvastatin | 28 timepoints up to day 10
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of Rosuvastatin and Atorvastatin | 28 timepoints up to day 10

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) of Rosuvastatin and Atorvastatin | 28 timepoints up to day 10
Terminal plasma half life (T-HALF) of Rosuvastatin and Atorvastatin | 28 timepoints up to day 10
Apparent total body clearance (CLT/F) of Rosuvastatin and Atorvastatin | 28 timepoints up to day 10
Safety based on results of physical examinations, vital sign measurements, ECGs, 24-hour telemetry, clinical laboratory tests, and physical measurements and will also include the incidence of AEs, SAEs and AEs leading to discontinuation | Up to day 10
  Adverse Event (AE)
  Serious Adverse Event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb